CLINICAL TRIAL: NCT00963885
Title: A Randomized, Partially-blind Study on the Safety, Tolerability and Effect on Virological Response of Treatment With the HCV Protease Inhibitor RO5190591 in Combination With Pegasys and Copegus, Versus Pegasys and Copegus Alone, in Treatment-Naïve Patients With Hepatitis C Genotype 1 Virus Infectio
Brief Title: A Study of RO5190591 (Danoprevir) in Combination With Pegasys and Copegus in Treatment-Naive Patients With Chronic Hepatitis C Genotype 1 Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV21075; 2009-009608-38
Record Dates: First submitted 2009-08-18; First posted 2009-08-24 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a; danoprevir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Part 1: Placebo (Placebo Comparator): Placebo in combination with standard doses of Pegasys and Copegus.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: Placebo
- Part 1: RO5190591 300mg po (Experimental): RO5190591 300mg po every 8 hours in combination with standard doses of Pegasys and Copegus.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO5190591 (Danoprevir)
- Part 1: RO5190591 600mg po (Experimental): RO5190591 600mg po every 12 hours in combination with standard doses of Pegasys and Copegus.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO5190591 (Danoprevir)
- Part 1: RO5190591 900mg po (Experimental): RO5190591 900mg po every 12 hours in combination with standard doses of Pegasys and Copegus.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO5190591 (Danoprevir)
- Part 2: Placebo (Placebo Comparator): If the safety and virological response data from Part 1 of the study are supportive, in Part 2 patients will be randomized to receive placebo in combination with standard doses of Pegasys and Copegus.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: Placebo
- Part 2: RO5190591 300mg po (Experimental): If the safety and virological response data from Part 1 of the study are supportive, in Part 2 patients will be randomized to receive RO5190591 300mg po every 8 hours or 600mg po every 12 hours or 900mg po every 12 hours in combination with standard doses of Pegasys and Copegus.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO5190591 (Danoprevir)

INTERVENTIONS:
Drug: Copegus — 1000 or 1200mg po daily for 24 or 48 weeks
Drug: Pegasys — 180micrograms sc weekly for 24 or 48 weeks
Drug: Placebo — po for 12 weeks
  Arms: Part 1: Placebo
Drug: Placebo — po for 24 weeks
  Arms: Part 2: Placebo
Drug: RO5190591 (Danoprevir) — 300mg po q8h for 12 weeks
  Arms: Part 1: RO5190591 300mg po
Drug: RO5190591 (Danoprevir) — 600mg po q12h for 12 weeks
  Arms: Part 1: RO5190591 600mg po
Drug: RO5190591 (Danoprevir) — 900mg po q12h for 12 weeks
  Arms: Part 1: RO5190591 900mg po
Drug: RO5190591 (Danoprevir) — 300mg po q8h or 600mg po q12h or 900po q12h for 24 weeks
  Arms: Part 2: RO5190591 300mg po

SUMMARY:
This 2 part study will evaluate the efficacy and safety of 12 and 24 weeks treatment with RO5190591 (danoprevir) in combination with Pegasys and Copegus, compared to Pegasys and Copegus alone, in treatment-naive patients with chronic hepatitis C genotype 1 virus infection.In Part 1 of the study, patients will be randomized to receive either 1) RO5190591 300mg po every 8 hours, 2) RO5190591 600mg po every 12 hours, 3) RO5190591 900mg po every 12 hours or 4) placebo, in combination with standard doses of Pegasys and Copegus. If the safety and virological response data from Part 1 of the study are supportive, in Part 2 patients will be randomized to receive either 1) RO5190591 300mg po every 8 hours or 600mg po every 12 hours or 900mg po every 12 hours or 2)placebo, in combination with standard doses of Pegasys and Copegus. The anticipated time on study treatment is 24-48 weeks, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic hepatitis C, genotype 1;
* treatment-naive.

Exclusion Criteria:

* liver cirrhosis and other forms of liver disease;
* HIV infection;
* hepatocellular cancer;
* cardiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2009-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Sustained virological response | 24 weeks after end of treatment

SECONDARY OUTCOMES:
Virological response over time | At 2- to 6-weekly intervals throughout study; at end of treatment; 12 weeks post-treatment
Adverse events; laboratory parameters | Throughout study, laboratory parameters every 2 to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (40):
- United States (23):
  - Phoenix, Arizona
  - Long Beach, California
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - Aurora, Colorado
  - Gainesville, Florida
  - Jacksonville, Florida
  - Orlando, Florida
  - Lombard, Illinois
  - New Orleans, Louisiana
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Manhasset, New York
  - New York, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Medford, Oregon
  - Lancaster, Pennsylvania
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Vancouver, Washington
  - Milwaukee, Wisconsin
- Australia (3):
  - Kingswood, New South Wales
  - Adelaide, South Australia
  - Heidelberg, Victoria
- Vienna, Austria
- Canada (6):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Ottawa, Ontario
  - Toronto, Ontario
- France (4):
  - Clichy
  - Marseille
  - Montpellier
  - Paris
- Germany (2):
  - Frankfurt am Main
  - Hamburg
- Napoli, Campania, Italy

REFERENCES:
- [Derived] Marcellin P, Cooper C, Balart L, Larrey D, Box T, Yoshida E, Lawitz E, Buggisch P, Ferenci P, Weltman M, Labriola-Tompkins E, Le Pogam S, Najera I, Thomas D, Hooper G, Shulman NS, Zhang Y, Navarro MT, Lim CY, Brunda M, Terrault NA, Yetzer ES. Randomized controlled trial of danoprevir plus peginterferon alfa-2a and ribavirin in treatment-naive patients with hepatitis C virus genotype 1 infection. Gastroenterology. 2013 Oct;145(4):790-800.e3. doi: 10.1053/j.gastro.2013.06.051. Epub 2013 Jun 26. PMID 23811112